CLINICAL TRIAL: NCT00709293
Title: Role of Intraoperative Thymoglobulin in Decreasing Ischemia-Reperfusion Injury in Pediatric Heart Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University of California, Los Angeles (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Juan Alejos, Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Thymoglobulin - Alejos
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Ischemia Reperfusion Injury; Heart Transplantation
Keywords: Ischemia Reperfusion Injury; Pediatric Heart Transplant; ATG; Induction Therapy
MeSH Terms: conditions — Reperfusion Injury | interventions — Antilymphocyte Serum; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Normal Saline
- 2 (Active Comparator)
  Interventions: Drug: Anti-Thymocyte Globulin

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin — Thymoglobulin (1.5 mg/kg body weight) will be infused through a peripheral intravenous line over a minimum of 6 hours. The infusion will be started at the time of donor visualization (once it is confirmed the transplant is proceeding). The peri-operative nurse or anesthesiologist will be responsible for drug infusion.
  Other Names: ATG
  Arms: 2
Drug: Normal Saline — Normal saline will be utilized as a placebo comparator. It will be infused in the same fashion as the Thymoglobulin in the intervention arm.
  Arms: 1

SUMMARY:
The restoration of normal blood flow following a period of ischemia may result in ischemia / reperfusion injury (I/RI), which is characterized by inflammation and oxidative damage to tissues. Varying degrees of I/RI occur upon reperfusion of a donor heart after cold storage. Medications containing antibodies against immune cells have been used for many years as powerful immunosuppressants. These medications, called polyclonal antibody preparations, are generally only used immediately following transplantation and/or to treat rejection. At our institution, one such antibody preparation (Thymoglobulin) is used in most pediatric heart transplant recipients for 3-5 days immediately after transplantation. Because standard immunosuppressive medications (called calcineurin inhibitors) are toxic to the kidneys, the use of Thymoglobulin allows us to delay the initiation of calcineurin inhibitors until the kidneys of completely recovered from the shock of the transplant surgery.

We hypothesize that Thymoglobulin may be beneficial in reducing the damage caused by I/RI. Thus, the present study seeks to evaluate the effectiveness of an intra-operative dose of Thymoglobulin (in addition to the standard doses post-operatively) at reducing the effects of I/RI. The study will be a double-bind placebo-controlled trial involving 20 subjects. Biologic markers for I/RI will be assessed at periodic intervals for six months post-transplantation. Subjects receiving intra-operative doses of Thymoglobulin will be compared to the controls in order to assess the effectiveness of intra-operative Thymoglobulin in ameliorating the effects of I/RI.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric population (ages 0-21 years)
* End-stage cardiac disease requiring heart transplantation
* Approval for listing by the UCLA Heart Transplant Committee

Exclusion Criteria:

* Prior documented Thymoglobulin allergy/adverse reaction
* History of or current diagnosis of lymphoma
* Documented lymphopenia
* Documented Thrombocytopenia
* Pregnancy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Alejos, MD, Principal Investigator — Department of Pediatrics, University of California Los Angeles
Locations (1):
- Mattel Children's Hospital at UCLA, Los Angeles, California, United States